CLINICAL TRIAL: NCT00477009
Title: A Randomized Controlled Trial of Effects From a Mandibular Advancement Device in Patients With Obstructive Sleep Apnea and Snoring
Brief Title: Effects From a Mandibular Repositioning Appliance in Patients With Obstructive Sleep Apnea and Snoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Marie Marklund, Associate professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: K2007-70X-20517-01-3; Dnr 07-032M
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Sleep Apnea Syndromes; Snoring; Disorders of Excessive Somnolence
Keywords: Sleep apnea syndromes; Snoring; Mandibular advancement; Activator appliances; Disorders of excessive somnolence; Blood pressure; Inflammation; Oxidative stress; Hormones; Markers of Metabolic Syndrome X
MeSH Terms: conditions — Sleep Apnea Syndromes; Snoring; Disorders of Excessive Somnolence; Inflammation | interventions — Orthodontic Appliances, Functional

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Adjustable mandibular repositioning appliance
  Interventions: Device: Mandibular repositioning appliance, adjustable
- 2 (Placebo Comparator): Placebo device in upper jaw
  Interventions: Device: Mandibular repositioning appliance, adjustable

INTERVENTIONS:
Device: Mandibular repositioning appliance, adjustable — Comparison between mandibular repositioning appliance for nightly use and a placebo device regarding effects on sleep apneas and daytime symptoms as well as blood pressure and markers of oxidative stress and sleepiness.
  Other Names: Herbst appliance

SUMMARY:
The purpose of this study is to evaluate effects from a mandibular repositioning appliance on obstructive sleep apneas, symptoms, blood pressure and markers of stress, inflammation and cardiovascular health in patients with mild to moderate obstructive sleep apnea/hypopnea syndrome and in patients with symptomatic snoring.

DETAILED DESCRIPTION:
Mandibular repositioning appliances for the treatment of snoring and sleep apneas are increasingly used over the world, although the number of prescriptions of this therapy varies between countries. The appliance widens the upper airways during sleep in order to reduce sleep-disordered breathing. The device is easy to use and has become popular among patients. Despite this, the evidence for effects of this treatment is not very strong and based on only a few studies. The aim of this study is therefore to test the hypothesis that a mandibular repositioning appliance reduces sleep apneas, daytime sleepiness and other sleep apnea symptoms and increases the quality of life in sleepy patients with mild to moderate obstructive sleep apnea and in patients with symptomatic snoring. Secondary outcomes include effects on headaches, blood pressure and markers of stress, inflammation, cardiovascular health and oxidative stress. At baseline and after 4 month's treatment, the patients will respond to questionnaires about symptoms and quality of life. They will undergo measurements of sleepiness, sleep apneas and blood pressure as well as sampling of saliva, urine and blood. Factors that predict a successful treatment outcome will be analyzed in order to more exactly clarify the indications for this treatment modality in a group of patients who have been suggested to benefit from mandibular repositioning appliances according to previous studies and reviews.

ELIGIBILITY:
Inclusion Criteria:

* Obstructive sleep apnea, apnea-hypopnea index of <30 with excessive daytime sleepiness
* Snoring with excessive daytime sleepiness, apnea-hypopnea index of <5
* Body mass index of <35

Exclusion Criteria:

* Unable to give informed consent
* Psychiatric disorders including dementia that may interfere with the study protocol
* Other concomitant diseases that demand acute, effective treatment of sleep apnea
* Pharyngeal soft tissue abnormalities
* Living to far away from the University Hospital
* Professional drivers
* Pregnancy
* Included in other studies
* Other sleep apnea treatments
* Severe craniomandibular disorders
* Acute or advanced periodontal disease
* Insufficient number of teeth

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2007-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Sleep apnea and sleep measured by polysomnography | Baseline and after 4 months
Daytime sleepiness and sleep apnea symptoms assessed in questionnaires and objective testing | Baseline and after 4 months
Quality of life | Baseline and after 4 months

SECONDARY OUTCOMES:
Headaches | Baseline and after 4 months
Blood pressure | Baseline and after 4 months
Vigilance | Baseline and after 4 months
Markers of stress | Baseline and after 4 months
Markers of inflammation | Baseline and after 4 months
Markers of cardiovascular health and oxidative stress | Baseline and after 4 months
Side-effects from the treatment | After 4 months treatment
Predictors of effects on symptoms and sleep apneas | After 4 months treatment

CONTACTS AND LOCATIONS:
Overall Officials: Marie Marklund, Principal Investigator — Umeå University
Locations (1):
- Depts of Respiratory Medicine and Orthodontics, Umeå University, Umeå, Sweden

REFERENCES:
- [Background] Marklund M, Stenlund H, Franklin KA. Mandibular advancement devices in 630 men and women with obstructive sleep apnea and snoring: tolerability and predictors of treatment success. Chest. 2004 Apr;125(4):1270-8. doi: 10.1378/chest.125.4.1270. PMID 15078734
- [Background] Lim J, Lasserson TJ, Fleetham J, Wright J. Oral appliances for obstructive sleep apnoea. Cochrane Database Syst Rev. 2006 Jan 25;2006(1):CD004435. doi: 10.1002/14651858.CD004435.pub3. PMID 16437488
- [Derived] Rietz H, Franklin KA, Carlberg B, Sahlin C, Marklund M. Nocturnal Blood Pressure Is Reduced by a Mandibular Advancement Device for Sleep Apnea in Women: Findings From Secondary Analyses of a Randomized Trial. J Am Heart Assoc. 2018 Jun 21;7(13):e008642. doi: 10.1161/JAHA.118.008642. PMID 29929990
- [Derived] Marklund M, Carlberg B, Forsgren L, Olsson T, Stenlund H, Franklin KA. Oral Appliance Therapy in Patients With Daytime Sleepiness and Snoring or Mild to Moderate Sleep Apnea: A Randomized Clinical Trial. JAMA Intern Med. 2015 Aug;175(8):1278-85. doi: 10.1001/jamainternmed.2015.2051. PMID 26030264